CLINICAL TRIAL: NCT02786992
Title: Adjuvant Use of Misoprostol and Oxytocin vs. Carbetocin for the Prevention of Post-partum Hemorrhage in Elective Cesarian Section
Brief Title: Misoprostol+Oxytocin vs. Carbetocin in CS
Acronym: CS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed S Sweed, MD, Dr, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AS1301
Record Dates: First submitted 2016-05-24; First posted 2016-06-01 (Estimated); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Cesarean Section
Keywords: Misoprostol; Oxytocin; Carbetocin; Prevention; Post-partum hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Misoprostol; Oxytocin; carbetocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Misoprostol + Oxytocin (Active Comparator): 400 ug sublingual misoprostol + 10 IU Oxytocin IVI
  Interventions: Drug: Misoprostol; Drug: Oxytocin; Drug: Placebo
- Carbetocin (Active Comparator): 100 ug Carbetocin IV
  Interventions: Drug: Carbetocin; Drug: Placebo

INTERVENTIONS:
Drug: Misoprostol
  Other Names: Mesotec; Mesotac
  Arms: Misoprostol + Oxytocin
Drug: Oxytocin
  Other Names: Syntocinon
  Arms: Misoprostol + Oxytocin
Drug: Carbetocin
  Other Names: Pabal
  Arms: Carbetocin
Drug: Placebo

SUMMARY:
This prospective randomized double-blind clinical trial will be conducted at Ain-Shams University Maternity Hospital, Cairo, Egypt. Patients eligible for elective lower segment cesarean section will be randomized to 2 groups. Group 1: will receive 400 ug misoprostol following + 10 IU oxytocin intravenous slowly after cord clamping. Group 2: will receive 100 ug carbetocin intravenous after cord clamping.

ELIGIBILITY:
Inclusion Criteria:

* Women with singleton pregnancy Women scheduled for elective CS full term (gestational age ≥37 weeks).

Exclusion Criteria:

* hypersensitivity to oxytocin, carbetocin or prostaglandins
* contraindication to prostaglandins (e.g. glaucoma)
* history of significant heart disease
* severe asthma
* epilepsy
* history or evidence of liver
* renal or vascular disease
* history of coagulopathy
* thrombocytopenia or anticoagulant therapy
* women with HELLP syndrome
* eclampsia
* women presenting by placental abruption
* contraindication to spinal anesthesia as carbetocin is licensed for use with regional anesthesia only.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Actual)
Dates: Start 2016-05; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
incidence of post-partum hemorrhage | 24 hours
amount of blood loss | 24 hours

SECONDARY OUTCOMES:
Number of participants needing extra uterotonic drug (10 IU oxytocin IVI) | 24 hours
  An experienced attendant (principal investigator) will assess the need of extra uterotonic drug (10 IU oxytocin IVI) if the uterus is atonic or if blood loss is more than 1000 ml.
Number of participants needing hemostatic surgical interventions | intra-operative
Hemoglobin deficit in gm/dl | 24 hours
  difference between pre-operative and 24 hours post-operative hemoglobin in gm/dl
APGAR score at 1 minute and 5 minutes | 1 minute and 5 minutes
Number of participants with NICU admission | 24 hours
Drug side effects | 24 hours
Time till resuming bowel habits | 24 hours
  Time of passing gas will be recorded how many hours post-operative
hematocrit deficit in % | 24 hours
  difference between pre-operative and 24 hours post-operative hematocrit in %

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt